CLINICAL TRIAL: NCT04282733
Title: Mindfulness Rounds Initiative - An 8-Week, Short Session, Mindfulness Based Protocol for On-Site Delivery of Stress Reduction Practices
Brief Title: Mindfulness Rounds Initiative - A Short Mindfulness-Based Program for A Busy Workplace
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No post-intervention survey completed
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jeffrey Zahn, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-1849
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Healthcare Practitioner Stress; Patient Satisfaction
Keywords: Mindfulness; Stress; pain scores; patient satisfaction; Perceived Stress Scale; MBSR
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The participants are staff on two hospital units tending to the same patient population with the same policies and protocols - postpartum patients. One unit will have the Mindfulness Rounds Initiative as the intervention, the other will not. Both units will be evaluated against each other, and against themselves in a pre-/post- design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Rounds (Experimental): Participants will be exposed to thrice weekly Mindfulness Rounds education on the Unit; participation in the actual sessions is voluntary.
  Interventions: Behavioral: Mindfulness Rounds
- Control (No Intervention): No intervention will take place on this Unit

INTERVENTIONS:
Behavioral: Mindfulness Rounds — Throughout the 8-week study period, a different mindfulness practice will be introduced weekly in 3 separate 15-minute live sessions. Posters describing the particular "practice of the week" will be placed around the Unit as visual reminders to encourage actual practice.
  Arms: Mindfulness Rounds

SUMMARY:
An 8 week course of mindfulness education and practices will be presented to all staff, patients, and visitors voluntarily attending the thrice weekly presentations. The goal is to reduce staff stress, improve communication, enhance patient satisfaction, and improve quality of care.

DETAILED DESCRIPTION:
"Mindfulness Rounds" Care-giver well-being is recognized as an important goal in decreasing burnout, increasing job satisfaction, and may have implications in improving quality of care and patient satisfaction. Mindfulness training is a well-studied tool used to enhance care-giver well-being. The impact of a Mindfulness training experience for caregivers, support staff, and patients and their families working together in a hospital unit on patient satisfaction has not been well studied, if at all. The researchers propose instituting a pilot program of Mindfulness Rounds on a given hospital unit and assessing the effect on employee well-being, patient satisfaction, and quality of care.

Introduction:

The physical and mental health of healthcare practitioners (HCPs) has become an area of attention and research in recent years as HCP burnout and suicide are now openly discussed concerns in medicine. Well-being education is now a required curricula component by the Accreditation Council for Graduate Medical Education (ACGME). Mindfulness is a technique and philosophical concept which has received significant attention in the medical literature as a tool for increasing HCP well-being.

Mindfulness describes the idea of maintaining a conscious presence in the present, of avoiding obsessing about the past or the future, and of continuously being aware of, and grateful for, the things we have in life as opposed to the things we don't. Mindfulness-Based Stress Reduction (MBSR) is one particular system, developed by Jon Kabat-Zinn over 30 years ago, which has been built into a well-structured certified training program for teaching mindfulness. Numerous studies have used MBSR or similar techniques to advance HCP psychologic well-being, and while some have investigated a variety of HCP training techniques to improve the patient experience, few have sought to explore a relationship between the impact of mindfulness training for HCP on patient satisfaction, quality of care outcomes, and HCP overall health. To the investigators' knowledge, no one has sought to bring mindfulness education to an entire hospital unit - physicians, nurses, support staff, as well as patients and their families wherever possible - with the goal of improving both HCP and the overall patient experience.

The researchers propose instituting a pilot program of Mindfulness Rounds on a given hospital unit and assessing the effect on employee well-being, patient satisfaction, and quality of care.

ELIGIBILITY:
Inclusion Criteria:

- Employees on the Units

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain scores | 1-3 months pre-intervention, 1-3 months post-intervention
  Patient pain scores are routinely collected by Nursing and entered into the electronic medical record (EMR). Full pain scale from 0-10, higher score indicates more pain.

SECONDARY OUTCOMES:
Discharge time | 1-3 months pre-intervention, 1-3 months post-intervention
  Duration from discharge order to discharge time.
Change in Narcotic usage | 1-3 months pre-intervention, 1-3 months post-intervention
  Aggregate total narcotics administered/patient hours on unit.
Change in Patient Satisfaction survey | 1-3 months pre-intervention, 1-3 months post-intervention
  Pres-Ganey survey to assess patient satisfaction. Pres-Ganey Survey: 24 item instrument, each item scored: very poor (score = 0), poor (25), fair (50), good (75) and very good (100). Full scale from 0 - 100, higher score indicates more satisfaction.
Change in Perceived Stress Scale (PSS) survey | Within 1 month prior to intervention, within one month post the intervention.
  This is a validated survey tool to assess an individual's perceived stress. Full scale range from 0 to 40, higher score indicates higher perceived stress.
Change in number of Staff sick days | 1-3 months pre-intervention, 1-3 months post-intervention
  Number of total staff sick days.
Change in number of staff injuries | 1-3 months pre-intervention, 1-3 months post-intervention
  Number of total staff injuries
Change in number of workers compensation claims | 1-3 months pre-intervention, 1-3 months post-intervention
  Number of total workers compensation claims
Change in number of discharges before noon | 1-3 months pre-intervention, 1-3 months post-intervention
  Number of discharges before noon as a hospital metric tracked for efficiency.
Change in Staff handwashing rates | 1-3 months pre-intervention, 1-3 months post-intervention
  Routinely tracked by anonymous observers

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zahn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No